CLINICAL TRIAL: NCT01587235
Title: A Multicenter, Open-label, 6 Week Study to Evaluate the Efficacy and Safety of Algorithm Based Intensive Treatment With Vytorin Versus Standard Treatment of Other Statins in Moderate, Moderately High and High Risk Patients.
Brief Title: A Study to Evaluate the Efficacy and Safety of Vytorin Versus Standard Treatment of Other Statins in Moderate, Moderately High and High Risk Participants (MK-0653A-406)
Acronym: VYCTORY
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653A-406
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vytorin (Experimental)
  Interventions: Drug: Ezetimibe/simvastatin
- Other Statin (Active Comparator)
  Interventions: Drug: Other Statin

INTERVENTIONS:
Drug: Ezetimibe/simvastatin — Algorithm based treatment using 10/10mg, 10/20mg and 10/40mg ezetimibe/simvastatin combination tablets orally once daily.
  Other Names: Vytorin
  Arms: Vytorin
Drug: Other Statin — Participants are prescribed a statin (any other than Vytorin) as per routine standard of care
  Arms: Other Statin

SUMMARY:
This study will evaluate and compare the effectiveness of MK-0653 (Vytorin) to current standard treatment with other statins for the treatment of dyslipidemia in moderate, moderately-high and high-risk participants.

ELIGIBILITY:
Inclusion Criteria:

* Low-density lipoprotein cholesterol (LDL-C) ≥100 mg/dL
* Either treatment naïve (no previous treatment with lipid-lowering medication) or if previously treated with lipid-lowering medication, must complete a wash-out 6 weeks prior to enrollment

Exclusion Criteria:

* LDL-C level ≥ 190 mg/dL
* Hypersensitivity or intolerance to Vytorin, ezetimibe or simvastatin
* Taking other lipid lowering agent except statins. (i.e. fenofibrate, niacin, ezetimibe, etc)
* Pregnant or breastfeeding, or expecting to conceive within the projected duration of the study
* Currently participating in or has previously participated in a study within 30 days
* Congestive heart failure defined by New York Heart Association (NYHA) Class III or IV within previous 6 months
* Uncontrolled cardiac arrhythmias or recent significant electrocardiogram (ECG) changes
* Unstable angina pectoris
* Myocardial infarction, coronary artery bypass surgery, or angioplasty within previous 3 months
* Unstable or severe peripheral artery disease within previous 3 months
* Uncontrolled hypertension (treated or untreated)
* Type 1 or Type 2 diabetes mellitus that is poorly controlled or recently diagnosed (within previous 3 months)
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins
* Serious cerebrovascular disorder (ischemic stroke or cerebral hemorrhage) within the previous 6 months
* Received treatment with systemic corticosteroids, any cyclical hormones

within previous 8 weeks

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Achieve Low-density Lipoprotein Cholesterol (LDL-C) goal (High-risk <100 mg/dL; Moderate-high and High risk <130 mg/dL) | Week 6

SECONDARY OUTCOMES:
Change in LDL-C level From Baseline | Baseline and Week 6
Number of High-risk Participants who Achieve an LDL-C < 70 mg/dL | Week 6
Change in Serum LDL From Baseline | Baseline and Week 6
Change in Total Cholesterol From Baseline | Baseline and Week 6
Change in High-density lipoprotein (HDL) From Baseline | Baseline and Week 6
Change in Serum Triglycerides (TG) From Baseline | Baseline and Week 6
Change in Serum Non-HDL From Baseline | Baseline and Week 6
Change in LDL-C/HDL-C Ratio From Baseline | Baseline and Week 6
Change in Apolipoprotein B (ApoB) From Baseline | Baseline and Week 6
Number of Participants who Achieve non-HDL-C goal (High-risk <100 mg/dL; Moderate-high and High risk <160 mg/dL)) | Week 6